CLINICAL TRIAL: NCT02724358
Title: Rg3 in Combination With TACE in Hepatocellular Carcinoma Patients With High Expression of Notch1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospital, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012ZX10002016008
Record Dates: First submitted 2016-03-28; First posted 2016-03-31 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma; TACE; Notch1; Rg3
Keywords: Carcinoma; Hepatocellular; Notch1
MeSH Terms: conditions — Carcinoma, Hepatocellular; Bicuspid Aortic Valve Disease; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- TACE (Experimental): iodized oil (5ml) + Pirarubicin (20mg)
  Interventions: Procedure: TACE
- Rg3 (Experimental): 20mg, BID, maintained though Month 12
  Interventions: Drug: Rg3
- TACE + Rg3 (Experimental): the combination of the treatments for the above two groups. Rg3 will be stopped on the day performing TACE.
  Interventions: Other: TACE + Rg3
- Control (Experimental): standard liver protective therapy
  Interventions: Procedure: protective therapy

INTERVENTIONS:
Procedure: TACE — iodized oil (5ml) + Pirarubicin (20mg)
  Other Names: Transcatheter Arterial Chemoembolization
  Arms: TACE
Drug: Rg3 — 20mg, BID, maintained though Month 12.
  Arms: Rg3
Other: TACE + Rg3
  Arms: TACE + Rg3
Procedure: protective therapy — standard liver protective therapy
  Arms: Control

SUMMARY:
In order to provide a new option for clinical anti-angiogenesis therapy in hepatoma, a randomized controlled study is planed to confirm the effect of Rg3 in combination with TACE on angiogenesis and tumor treatment in advanced hepatocellular carcinoma patients with high expression of Notch1.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed hepatocellular carcinoma.
2. High expression of Notch1 in tumor tissues.

Exclusion Criteria:

no pathological evidence of HCC

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 3 years
Time to progression | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China